CLINICAL TRIAL: NCT03326232
Title: Real-time Continuous Glucose Monitoring for the Treatment of Gestational Diabetes: a Randomized Trial
Brief Title: Real-time Continuous Glucose Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-07-FB-0181
Record Dates: First submitted 2017-10-25; First posted 2017-10-31 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blinded continuous glucose monitoring (Experimental): The blinded CGM group will be using the Medtronic iPro2 system (Enlite sensor + iPro2 transmitter).
  Interventions: Device: Continuous glucose monitoring
- Real time continuous glucose monitoring (Experimental): The real-time CGM group will be using the 530g system (inactivated 530g insulin pump (no insulin used, only used as display for CGM), Enlite sensor, MiniLink transmitter)
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — The blinded CGM group will be using the Medtronic iPro2 system (Enlite sensor + iPro2 transmitter). The real-time CGM group will be using the 530g system (inactivated 530g insulin pump (no insulin used, only used as display for CGM), Enlite sensor, MiniLink transmitter)

SUMMARY:
Gestational diabetes (GDM) is a condition of carbohydrate intolerance with onset or first recognition in pregnancy. The prevalence of GDM is as high as 25% in some populations and continues to rise with the increase in obesity and type-2 diabetes. GDM places the pregnancy at great risk to both the mother and the neonate. Recent studies have proven that interventions including dietary and medications lower the risk to the pregnancy. Both the American College of Obstetrics and Gynecology (ACOG) and the American Diabetes Association (ADA) recommend dietary interventions with daily glucose monitoring as the initial treatment of choice. Meanwhile, outside of pregnancy, promising new technologies such as continuous glucose monitors (CGM) are revolutionizing diabetic care. The investigators seek to determine if the constant feedback of a real-time CGM system would improve glycemic control compared to traditional management in GDM

DETAILED DESCRIPTION:
The investigators' proposed study will add new information to the emerging use of CGM in pregnant women with GDM. First, most studies only use CGM for 48 - 72hours at a time, while the investigators will be using CGM for 7 day intervals. Both groups will use the same Enlite sensor (Medtronic). The blinded CGM group will be using the Medtronic iPro2 system (Enlite sensor + transmitter). The real-time CGM group will be using the 530g system (iPro2 (Enlite sensor + transmitter) + inactivated 530g pump set only to display glucose values, no insulin will be administered). This CGM system has been FDA approved to for up to 7 days between sensor changes.26,27 Second, no previous study has used real time CGM in pregnant patients with GDM in the US. The investigators will be the first to describe the use of this technology in this patient population. Third, most of these trials have been performed on populations that are not representative of the investigators' patient population at EVMS. This will be the largest US study of CGM in GDM. Fourth wearable medical and fitness technology is already popular, but as both the technology and the demand continues to grow, it will become the future of diabetes management. Studies have already shown that real time CGM is an effective educational and motivational tool in type-1 and type-2 DM.28,29

ELIGIBILITY:
Inclusion Criteria:

* maternal age 18 to 45
* singleton gestation
* gestational age less than 32 weeks gestation at study inclusion
* BMI less than 45
* 50g glucose challenge greater than 135 mg/dL
* 100 g 3 hr oral glucose tolerance test greater than 2 abnormal values using the Carpenter Coustan cut offs (fasting greater than 95 mg/dL, 1 hr greater than 180 mg/dL, 2 hr greater than 155 mg/dL, 3 hr greater than 140 mg/dL)
* attended the maternal-fetal medicine diabetes education class

Exclusion Criteria:

* maternal age less than18 or greater than 45
* multifetal gestation
* gestational age greater than 32 weeks study inclusion
* BMI greater than 45
* pregestational diabetes
* gestational diabetes diagnosed before 24 weeks
* did not attend the diabetes education class
* known fetal anomaly
* known fetal aneuploidy
* required ongoing treatment with medications that can exacerbate hyperglycemia (steroids, hydroxyprogesterone caproate injections (Makena), highly active antiretroviral therapy HIV medications)
* learning disability
* concern for non compliance with medical care
* imminent preterm delivery due to maternal disease or fetal conditions
* is not willing to wear CGM

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females with gestational diabetes
Enrollment: 40 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Mean blood glucose (mg/dL) | week 1 vs. week 4
  Mean blood glucose (mg/dL) in the real-time CGM group compared to self-monitoring of blood glucose (SMBG) group during the 4th week of study from data collected on the 6 day of CGM use during that week.

SECONDARY OUTCOMES:
Failed dietary therapy | week 1 vs. week 4
  Failed dietary therapy (started on medication),
Time spent in normoglycemia | week 1 vs. week 4
  Time spent in normoglycemia (min/day)
Time spent in hypoglycemia | week 1 vs. week 4
  Time spent in hypoglycemia (min/day)
BMI at time of delivery | BMI at time of delivery
  BMI at time of delivery (kg/m2)
Gestational hypertension | enrollement vs delivery.
  Gestational hypertension (defined as systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mmg Hg, on 2 occasions at least 4 hrs apart
Preeclampsia | enrollement vs delivery.
  Preeclampsia (defined as gestational hypertension plus either new-onset proteinuria (> 300 mg/24 2hrs, protein:creatinine > 0.3 mg/dL), thrombocytopenia (platelet count < 100,000/uL), elevated Aspartate aminotransferase or alanine aminotransferase (> 2x upper limit of normal), renal insufficiency (serum creatinine > 1.1 mg/dL or an unexplained doubling of creatinine), pulmonary edema, or cerebral or visual symptoms
HbA1C values | HbA1C values week 1 compared to week 4 (%)
  HbA1C values (%)
Polyhydramnios | Through study completion, an average of 9 months
  Polyhydramnios (MVP > 8 cm at any point in the pregnancy)
Cesarean delivery | Delivery
  Cesarean delivery (w/ indication: macrosomia, malpresentation, failed induction, fetal distress, failed trial of labor after cesarean, scheduled repeat, other)
Induction of labor | Delivery
  Induction of labor (w/ indication)
Operative vaginal delivery | Delivery
  Operative vaginal delivery (yes/no) and type (forceps/vacuum)
Shoulder dystocia | Delivery
  Shoulder dystocia (diagnosed clinically)
Fetal macrosomia | Most recent ultrasound before delivery
  Fetal macrosomia (> 4,000g at 38 wk u/s)
3rd or 4th degree perineal laceration | Delivery
  3rd or 4th degree perineal laceration at time of delivery
Gestational age at delivery | Delivery
  Gestational age at delivery (weeks, days)
Preterm delivery | Delivery
  Preterm delivery (< 37 weeks gestational age at birth)
Birth weight | Delivery
  Birth weight (grams)
Perinatal morbidity composite outcome | Delivery
  * Hypoglycemia (yes/no): < 2 hrs after birth and before feeding, defined as < 35mg/dL
  * Hyperbilirubinemia (yes/no): collected 16-36 hrs after birth, defined as > 95% for any given point after birth requiring phototherapy according to American Academy of Pediatrics guidelines
  * Birth trauma (yes/no): brachial plexus injury or clavicular, humeral, or skull fracture
  * Intrauterine fetal demise or neonatal death (yes/no): prior to hospital discharge
Large for gestational age | Delivery
  Large for gestational age (yes/no): defined as birth weight > 90%
Small for gestational age | Delivery
  Small for gestational age (yes/no): defined as birth weight < 10%
Admission to neonatal intensive care unit | Delivery
  Admission to neonatal intensive care unit (yes/no) and length of neonatal intensive care unit stay (days)
Respiratory distress syndrome | Delivery
  Respiratory distress syndrome (defined as need to supplemental oxygen > 4 hrs after birth)

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Mlynarczyk, MD, PhD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Do not plan to share.

REFERENCES:
- [Background] Practice Bulletin No. 137: Gestational diabetes mellitus. Obstet Gynecol. 2013 Aug;122(2 Pt 1):406-416. doi: 10.1097/01.AOG.0000433006.09219.f1. PMID 23969827
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for gestational diabetes mellitus: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 18;160(6):414-20. doi: 10.7326/M13-2905. PMID 24424622
- [Background] Correa A, Bardenheier B, Elixhauser A, Geiss LS, Gregg E. Trends in prevalence of diabetes among delivery hospitalizations, United States, 1993-2009. Matern Child Health J. 2015 Mar;19(3):635-42. doi: 10.1007/s10995-014-1553-5. PMID 24996952
- [Background] England LJ, Dietz PM, Njoroge T, Callaghan WM, Bruce C, Buus RM, Williamson DF. Preventing type 2 diabetes: public health implications for women with a history of gestational diabetes mellitus. Am J Obstet Gynecol. 2009 Apr;200(4):365.e1-8. doi: 10.1016/j.ajog.2008.06.031. Epub 2008 Aug 8. PMID 18691691
- [Background] Boney CM, Verma A, Tucker R, Vohr BR. Metabolic syndrome in childhood: association with birth weight, maternal obesity, and gestational diabetes mellitus. Pediatrics. 2005 Mar;115(3):e290-6. doi: 10.1542/peds.2004-1808. PMID 15741354
- [Background] Malcolm JC, Lawson ML, Gaboury I, Lough G, Keely E. Glucose tolerance of offspring of mother with gestational diabetes mellitus in a low-risk population. Diabet Med. 2006 May;23(5):565-70. doi: 10.1111/j.1464-5491.2006.01840.x. PMID 16681566
- [Background] Gillman MW, Rifas-Shiman S, Berkey CS, Field AE, Colditz GA. Maternal gestational diabetes, birth weight, and adolescent obesity. Pediatrics. 2003 Mar;111(3):e221-6. doi: 10.1542/peds.111.3.e221. PMID 12612275
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Background] Hartling L, Dryden DM, Guthrie A, Muise M, Vandermeer B, Donovan L. Benefits and harms of treating gestational diabetes mellitus: a systematic review and meta-analysis for the U.S. Preventive Services Task Force and the National Institutes of Health Office of Medical Applications of Research. Ann Intern Med. 2013 Jul 16;159(2):123-9. doi: 10.7326/0003-4819-159-2-201307160-00661. PMID 23712381
- [Background] Klonoff DC. Continuous glucose monitoring: roadmap for 21st century diabetes therapy. Diabetes Care. 2005 May;28(5):1231-9. doi: 10.2337/diacare.28.5.1231. No abstract available. PMID 15855600
- [Background] Mastrototaro J, Shin J, Marcus A, Sulur G; STAR 1 Clinical Trial Investigators. The accuracy and efficacy of real-time continuous glucose monitoring sensor in patients with type 1 diabetes. Diabetes Technol Ther. 2008 Oct;10(5):385-90. doi: 10.1089/dia.2007.0291. PMID 18715215
- [Background] Kestila KK, Ekblad UU, Ronnemaa T. Continuous glucose monitoring versus self-monitoring of blood glucose in the treatment of gestational diabetes mellitus. Diabetes Res Clin Pract. 2007 Aug;77(2):174-9. doi: 10.1016/j.diabres.2006.12.012. Epub 2007 Jan 16. PMID 17234297
- [Background] Murphy HR, Rayman G, Lewis K, Kelly S, Johal B, Duffield K, Fowler D, Campbell PJ, Temple RC. Effectiveness of continuous glucose monitoring in pregnant women with diabetes: randomised clinical trial. BMJ. 2008 Sep 25;337:a1680. doi: 10.1136/bmj.a1680. PMID 18818254
- [Background] Moy FM, Ray A, Buckley BS. Techniques of monitoring blood glucose during pregnancy for women with pre-existing diabetes. Cochrane Database Syst Rev. 2014 Apr 30;(4):CD009613. doi: 10.1002/14651858.CD009613.pub2. PMID 24782359
- [Background] de Veciana M, Major CA, Morgan MA, Asrat T, Toohey JS, Lien JM, Evans AT. Postprandial versus preprandial blood glucose monitoring in women with gestational diabetes mellitus requiring insulin therapy. N Engl J Med. 1995 Nov 9;333(19):1237-41. doi: 10.1056/NEJM199511093331901. PMID 7565999
- [Background] Porter H, Lookinland S, Belfort MA. Evaluation of a new real-time blood continuous glucose monitoring system in pregnant women without gestational diabetes. A pilot study. J Perinat Neonatal Nurs. 2004 Apr-Jun;18(2):93-102. doi: 10.1097/00005237-200404000-00004. PMID 15214248
- [Background] McLachlan K, Jenkins A, O'Neal D. The role of continuous glucose monitoring in clinical decision-making in diabetes in pregnancy. Aust N Z J Obstet Gynaecol. 2007 Jun;47(3):186-90. doi: 10.1111/j.1479-828X.2007.00716.x. PMID 17550484
- [Background] Yu F, Lv L, Liang Z, Wang Y, Wen J, Lin X, Zhou Y, Mai C, Niu J. Continuous glucose monitoring effects on maternal glycemic control and pregnancy outcomes in patients with gestational diabetes mellitus: a prospective cohort study. J Clin Endocrinol Metab. 2014 Dec;99(12):4674-82. doi: 10.1210/jc.2013-4332. PMID 25057872
- [Background] Alfadhli E, Osman E, Basri T. Use of a real time continuous glucose monitoring system as an educational tool for patients with gestational diabetes. Diabetol Metab Syndr. 2016 Jul 26;8:48. doi: 10.1186/s13098-016-0161-5. eCollection 2016. PMID 27468313
- [Background] Glowinska-Olszewska B, Tobiaszewska M, Luczynski W, Bossowski A. Monthly use of a real-time continuous glucose monitoring system as an educational and motivational tool for poorly controlled type 1 diabetes adolescents. Adv Med Sci. 2013;58(2):344-52. doi: 10.2478/ams-2013-0024. PMID 23917476

DOCUMENTS (1):
  • Study Protocol (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT03326232/Prot_000.pdf